CLINICAL TRIAL: NCT06019819
Title: Effects of 4 Weeks Postural Correction Exercises in Reducing Forward Head Posture in Children Carrying Heavy Bag Packs
Brief Title: Effects of Postural Correction Exercises in Reducing Forward Head Posture in Children Carrying Heavy Bag Packs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MSPT/01689 Sidrah Sufian
Record Dates: First submitted 2023-08-26; First posted 2023-08-31 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Postural Kyphosis
Keywords: forward head posture; posture correction exercises; strength training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General training group A (Active Comparator): Perform general physical training activities conducted in schools including upper limb forward elevation, lateral elevation, touching toes in standing and cervical range of motion, strengthening exercise will be performed.
  Interventions: Other: strengthening exercise
- Postural correction exercises group B (Experimental): Chin Tuck, Strengthening shoulder retractors, Stretching sternocleidomastoiD, Pectorals stretch
  .
  Interventions: Other: Postural correction exercises

INTERVENTIONS:
Other: strengthening exercise — Perform general physical training activities conducted in schools including upper limb forward elevation, lateral elevation, touching toes in standing and cervical range of motion, strengthening exercise will be performed for 3days a week for 4 weeks.
  Arms: General training group A
Other: Postural correction exercises — Chin Tuck, Strengthening shoulder retractors, Stretching sternocleidomastoiD, Pectorals stretch For strengthening exercises 3 sets of 10 repetitions were performed with 6 seconds rest period between each set and a hold of 6 seconds. Stretching exercises will be performed in 3 sets of 10 repetitions ,30 seconds hold and 30 seconds rest period between each exercise. The exercises were performed 3days a week for 4 weeks.
  Arms: Postural correction exercises group B

SUMMARY:
This study aims to investigate the effectiveness of a 4-week postural correction exercise program in reducing FHP in children carrying heavy backpacks to school. This study's findings could have significant implications for preventing musculoskeletal problems associated with FHP. Furthermore, the study's findings could inform healthcare professionals and educators about the importance of promoting healthy postures among children and adolescents to prevent long-term musculoskeletal problems. This is an experimental study. Subjects will be divided into two groups. Group A (control group) and group B (experimental group).fun activities will be performed by experimental group under the supervision of the therapist.

DETAILED DESCRIPTION:
Regular use of heavy school bags and inappropriate carrying methods can put children at the risk of musculoskeletal problems and changes the body posture. It is imperative to note that carrying a backpack more than the recommended weight limit poses a twofold hazard, particularly to children and adolescents who are undergoing neuromusculoskeletal development and growth. Hence, it is crucial to ensure that the backpack's weight does not exceed 10-15% of the child or adolescent's body weight. Overreaching this weight limit may result in posterior displacement of the center of gravity, thereby engendering augmented strain on the neck and back muscles. Such effects are commonly linked with spinal column pathologies and reduced lung volume.One of the most prevalent types of postural anomaly is called "forward head posture" (FHP), and it is typically characterized by the head being anterior to the body's vertical line gravity point. Chronic FHP issues develop from an excessive load being placed on the joint and muscle when cervical muscular imbalances brought on by postural misalignment are left untreated. Both an upper cervical extension and a lower cervical flexion define forward head position. These modifications in the cervical region could result in long-term bad head posture, which could cause "upper crossed syndrome" or other musculoskeletal disorders. Additionally, neck and shoulder pain are common complaints among FHPs patients . Numerous studies have shown that carrying a backpack that is 7.5% of or more of your body weight (BW) causes postural compensations. The increased weight of the backpack correlates with higher FHP, trunk flexion, spinal asymmetry, and tensile forces in the intervertebral discs under static settings

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Children who carry heavy backpacks to school (more than 10% of their body weight)
* Forward head posture, defined as a craniovertebral angle of less than 50 degrees.
* Willing to participate in the study.
* Consent obtained from parents or legal guardians

Exclusion Criteria:

* Cervical spine fracture or neurological disorder.
* Scoliosis or torticollis.
* Joint hypermobility or recent surgery . Prior history of physical therapy treatment for forward head posture in the past six months

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Forward head posture analysis app | 4 weeks
  Changes form the Baseline will be measured. This Forward head posture analysis app can be used to assess the forward head posture using visual analysis through camera. the angle of the cervical spine was measured in the side view through pictures.

SECONDARY OUTCOMES:
numeric pain rating scale | 4th week
  Changes form the Baseline will be measured. It measured the neck pain with 11 points, 0 showing min and 10 showing max pain

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Private and Public Schools, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No